CLINICAL TRIAL: NCT00540085
Title: Pharmacodynamic Trial on Rocuronium in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Lars S. Rasmussen, Department of Anaesthesia, HOC, Copenhagen University Hospital, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2007-003005-27; H-B-2007-038
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Rocuronium dosed after ideal body weight
  Interventions: Drug: Rocuronium
- B (Active Comparator): Rocuronium dosed after corrected body weight 20%
  Interventions: Drug: Rocuronium
- C (Active Comparator): Rocuronium dosed after corrected body weight 40%
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — 0.6 mg/kg given intravenously before intubation
  Other Names: Esmeron (R)

SUMMARY:
Aim: To optimize the use of rocuronium (a neuromuscular blocking agent) in obese patients undergoing gastric bypass or gastric banding.

Background: During general anaesthesia, a neuromuscular blocking agent is needed to allow surgery and airway management. Optimal dosing is important in order to avoid inadequately muscle relaxation, but also to avoid overdosage, which can result in prolonged anaesthesia and respiratory complications.

Main hypothesis: Rocuronium dosed according to ideal body weight results in shorter duration of action compared to rocuronium dosed according to corrected body weight without prolonged onset time or compromised airway management or surgical demands for muscle relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Elective laparoscopic gastric banding or gastric bypass.

Exclusion Criteria:

* Expected difficult endotracheal intubation based on anatomic or pathologic findings or history.
* Known or suspected neuromuscular disease, known to affect the neuromuscular blockade.
* Severely impaired renal or hepatic function, as evaluated by the investigator.
* Known or suspected allergy to drugs used in the trial.
* Daily or expected use during the trial of the following drugs, known to affect neuromuscular transmission: Inhalational anaesthetics, magnesiumsalts, clindamycin, polymyxins and aminoglycosides (gentamicin, neomycin, netilmicin, streptomycin og tobramycin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Duration of action, defined as: Time to reappearance of T4. | 1 day

SECONDARY OUTCOMES:
Complete duration of action, defined as: Time to TOF-ratio = 0.9 | 1 day
Onset time | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lars S Rasmussen, MD, DMSc, Study Chair — Department of anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Denmark; Christian S Meyhoff, MD, PhD, Principal Investigator — Department of anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Denmark; Casper Claudius, MD, PhD, Study Director — Department of anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Denmark; Jørgen Viby-Mogensen, Prof., DMSc, Study Director — Department of anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Denmark; Jørgen Lund, MD, Study Director — Department of anaesthesia, Privathospitalet Hamlet A/S, Denmark; Morten Jenstrup, MD, Study Director — Department of anaesthesia, Privathospitalet Hamlet A/S, Denmark; Anne Marie Sørensen, MD, PhD, Study Director — Department of anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Department of anaesthesia, Privathospitalet Hamlet A/S, Copenhagen, Denmark

REFERENCES:
- [Result] Meyhoff CS, Lund J, Jenstrup MT, Claudius C, Sorensen AM, Viby-Mogensen J, Rasmussen LS. Should dosing of rocuronium in obese patients be based on ideal or corrected body weight? Anesth Analg. 2009 Sep;109(3):787-92. doi: 10.1213/ane.0b013e3181b0826a. PMID 19690247